CLINICAL TRIAL: NCT04116294
Title: Using a Computer-assisted Prescription to Decrease Inappropriate Use of Plain Abdominal Radiography in Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christophe Fehlmann (Other)
Responsible Party: Sponsor-Investigator, Christophe Fehlmann, Junior attending, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-02142
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Plain Abdominal Radiography

STUDY DESIGN:
Intervention Model Description: Before after. During the before period, standard of care. During the after period, computer-assisted prescription for plain abdominal radiography (reminding the indication for this procedure).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before (No Intervention): Standard of care for informatic prescription.
- After (Active Comparator): Computer-assisted prescription for radiological procedure
  Interventions: Other: Computer-assisted prescription

INTERVENTIONS:
Other: Computer-assisted prescription — The intervention is based on a computer-assisted prescription: when a PAR will be ordered, an alert will arise and explain the recognized indications for this examination and ask a confirmation for the prescription. This is a non-blocking system: physicians will be able to prescribe PAR even if the PAR is not appropriate.
  Arms: After

SUMMARY:
The aim of this study is to assess whether a computer-assisted prescription allows a reduction of the overall number of inappropriate PAR in emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 or more with a PAR.

Exclusion Criteria:

* Refusal to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of plain abdominal radiopraphy (PAR) with an inappropriate indication | Same ED consultation (or max 24 hours)
  4 indications are considered as appropriate : (1) foreign body suspicion, (2) checking after contrast injection, (3) catheter checking and (4) follow-up of urolithiasis. Order for PAR will be independantly reviewed by blinded assessors.

SECONDARY OUTCOMES:
Incidence of additional radiological examination (CT, US, IRM) after the PAR | Same ED consultation (or max 24 hours)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Hôpitaux Universitaires de Geneve, Geneva
  - Hôpital de La Tour, Meyrin

IPD SHARING:
Plan to Share IPD: No